CLINICAL TRIAL: NCT01845688
Title: Efficacy and Safety Evaluation of QingReMoShen Granule in the Treatment of Idiopathic Membranous Nephropathy : A Randomized Double-Blind Controlled Clinical Study
Brief Title: Clinical Study of QingReMoShen Granule to Treat Idiopathic Membranous Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: wanglin (Other)
Responsible Party: Sponsor-Investigator, wanglin, Deputy director of Physicians, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShanghaiSTCSM-2011; 11DZ1972703 (Other Grant/Funding Number: Shanghai Science and Technology Commission)
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: Idiopathic Membranous Nephropathy; Traditional Chinese Medicine; Randomized Control Trial
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Losartan Tablets & QingReMoShen Granule (Experimental): Losartan Tablets: 50mg, qd, po. QingReMoShen Granule: 12g, tid, po.
  Interventions: Drug: Losartan Tablets & QingReMoShen Granule
- Losartan Tablets & Placebo Granule (Placebo Comparator): Losartan Tablets: 50mg, qd, po. Placebo Granule: 12g, tid, po.
  Interventions: Drug: Losartan Tablets & Placebo Granule

INTERVENTIONS:
Drug: Losartan Tablets & QingReMoShen Granule
  Arms: Losartan Tablets & QingReMoShen Granule
Drug: Losartan Tablets & Placebo Granule
  Arms: Losartan Tablets & Placebo Granule

SUMMARY:
The purpose of this study is to evaluate the clinical safety and efficacy of QingReMoShen Granule to treat idiopathic membranous nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Women and men who had a clinic and biopsy-proven idiopathic membranous nephropathy;
* 6.0g≥24 hour urinary protein≥1.0g;
* serum albumin concentration≥26g/L;
* Chronic Kidney Disease (CKD)≤3 stage (eGFR>30ml/min/1.73m2 MDRD);
* Willing to participate in the trial and signed an informed consent.

Exclusion Criteria:

* Secondary membranous nephropathy;
* Patients with one of the following circumstances- malignant tumors or malignancy, HIV infection, a history of mental illness, any serious systemic infection, serious gastrointestinal diseases, circulating hepatitis B surface antigens positive or persistent abnormal serum transaminase, abnormal glucose metabolism or diabetes mellitus;
* Pregnant and lactating women;
* Undergoing other clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-11; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
24-hour urine protein | At the 24thweek

SECONDARY OUTCOMES:
serum albumin concentration | At the 24thweek
eGFR | At the 24thweek
Alanine transaminase | At the 24thweek

OTHER OUTCOMES:
T-cell classification | At the 24thweek
  Detecting by flow cytometry method

CONTACTS AND LOCATIONS:
Overall Officials: Lin Wang, PHD,MD, Study Director — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952